CLINICAL TRIAL: NCT04250831
Title: Impact of Dietary Fibre and Chromium Picolinate on Satiety, Satiation, Weight Loss and Gut Microbiome Composition in Overweight and Obese Women
Brief Title: Dietary Fibre and Chromium Picolinate Efficacy in Overweight and Obese Women
Acronym: DFCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, PI, University of Roehampton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSC 18/238
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Overweight; Obesity
Keywords: hormones; microbiota; mood; hunger; weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — oligofructose

STUDY DESIGN:
Intervention Model Description: Single group, prospective, open label pilot human intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucomannan, oligofructose and chromium mixture (Experimental): Agglomerated glucomannan, oligofructose and chromium mixture as the functional ingredient in a calorie
  Interventions: Dietary Supplement: agglomerated glucomannan, oligofructose and chromium mixture

INTERVENTIONS:
Dietary Supplement: agglomerated glucomannan, oligofructose and chromium mixture — Participants visited the University of Roehampton on three separate occasions: visit 1 (screening), visit 2 (baseline), and visit 3 (end of the trial) in total over a period of 4-weeks. During the 4-week study period, participants were instructed to replace breakfast and lunch with a shake (206 kcal/shake) each delivering 3g of the active ingredient (Mix: agglomerated glucomannan, oligofructose and chromium picolinate), and one snack bar each delivering 1.5g of the active ingredient (112 kcal/bar) in between breakfast and lunch, and lunch and dinner following by a selection of healthy dinner according to standard nutritional guidance not exceeding 1500 kcal/day. All subjects were instructed to prepare shakes by using a shaker or blender by mixing all ingredients with 200 ml of water. Participants were also instructed to consume all shakes and bars with an extra 200 ml glass of water throughout the study period.

SUMMARY:
Obesity is one of the greatest causes of preventable morbidity and mortality worldwide with the main treatments requiring significant changes to lifestyle, particularly dieting and physical exercise. Glucomannan is a dietary fibre that expands in the stomach, creating the feeling of fulness, while chromium can regulate insulin response.

DETAILED DESCRIPTION:
The aim of this pilot study was to investigate the effect of agglomerated glucomannan, oligofructose and chromium, as part of a calorie restricted diet plan, on weight loss, satiety, satiation, mood and gut microbiome composition in a human intervention study.

ELIGIBILITY:
Inclusion Criteria:

* healthy female
* aged 18-65 years
* with a BMI between 25 and 35 kg/m2
* not dieting within the previous four months
* not having lost > 5% body weight in the previous year
* not having increased physical activity levels in the past 2-4 weeks
* intending to modify them during the study
* able to eat most everyday foods

Exclusion Criteria:

* BMI < 25 kg/m2
* > 35 kg/m2
* significant health problems
* taking any medication or supplements known to affect appetite
* weight within the past month and/or during the study
* pregnant, planning to become pregnant or breastfeeding
* history of anaphylaxis to food
* known allergies or intolerance to foods and/or to the study materials or any of their stated ingredients.
* Volunteers who were on specific food avoidance diets
* with abnormal eating behaviour
* receiving systemic or local treatment likely to interfere with the evaluation of the study parameters
* smokers and those who have recently ceased smoking
* Volunteers who work in appetite or feeding related areas volunteers who participated in another experimental study or receipt of

Ages: 22 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Weight loss changes from the baseline to 4 weeks intervention | To test, in humans, changes in body weight from the baseline to 4 weeks intervention
  The body mass was measured to the nearest 0.1 kg using a digital balance scale (Seca 707, Seca Corporation, Hamburg, Germany)
Body mass index changes from the baseline to 4 weeks intervention | To test, in humans, changes in body mass index (calculated in Kg/m^2) from the baseline to 4 weeks intervention
  Body mass index was determined as weight divided by height squared (kg/m^2)
Blood pressure changes from the baseline to 4 weeks intervention | To test, in humans, changes in blood pressure (calculated in mm/Hg) from the baseline to 4 weeks intervention
  Blood pressure was measured using a digital blood pressure monitor (Nissei, model DS-1902, Japan Precision Instruments, Inc., Gunma, Japan).
Body composition changes from baseline to 4 weeks intervention | To test, in humans, changes in body fat percentage (calculated in %) from the baseline to 4 weeks intervention
  Body fat percentage was assessed after a 12-hour water-only fast by bioelectrical impedance analysis (BIA) method, using a Tanita BC-418 MA Segmental Body Composition Analyser, which incorporates eight tactile electrodes (Tanita Corporation, Tokyo, Japan).
Waist circumference changes from baseline to 4 weeks intervention | To test, in humans, changes in waist circumference (calculated in cm) from the baseline to 4 weeks intervention
  Waist was assessed using anthropometric tape (Seca 201, Hamburg, Germany) over light clothing to the nearest 0.1 centimetre while the subjects were in the standing position at the end of gentle expiration. The waist circumference was measured at the mid-point between the lowest rib margin and anterior superior iliac crest and hip circumference was measured at the maximum protuberance of the buttocks, and the waist-to-hip ratio was calculated by dividing waist circumference by hip circumference.
Resting metabolic rate changes from baseline to 4 weeks intervention | To test, in humans, changes in resting metabolic rate (calculated Kcal) from the baseline to 4 weeks intervention
  Resting metabolic rate (RMR) before and at the end of the 4-week intervention was determined by indirect calorimetry using the breath-by-breath system of recording (Cortex MetaLyzer 3B device).

SECONDARY OUTCOMES:
DNA Gut microbiome diversity changes from baseline to 4 weeks intervention | To test, in humans, changes in the faecal microbiota composition and microbial activity of the volunteers using DNA profiling in faeces from the baseline to 4 weeks
  Sequencing was performed on an Illumina MiSeq desktop sequencer using the MiSeq Reagent Kit V2 (Illumina, San Diego). The significance in the abundance of the relevant taxa were validated by Wilcoxon signed-rank tests (16s rRNA sequencing using Illumina MiSeq Platform and QIIME data analysis software).
Hunger, mood and cravings changes from baseline to 4 weeks intervention | To test, in humans, changes in hunger, mood and cravings (questionnaire based analysis) from the baseline to 4 weeks intervention
  Changes in hunger, mood and craving was determined via Control of Eating Questionnaire (CoEQ) comprised of twenty items to assess the intensity and type of food cravings each participant experienced over the previous 7 days, as well as subjective sensations of appetite and mood. Responses were recorded using the visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: ADELE COSTABILE, Dr, Study Director — Roehampton University
Locations (1):
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom